CLINICAL TRIAL: NCT05281952
Title: Medico-economic Evaluation of Management Strategies for Severe Epistaxis
Acronym: EPICOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/19-0550; 2020-A02824-35 (Other: ID-RCB)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Epistaxis
Keywords: Severe epistaxis; endoscopic ligation; Supra-selective embolization
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Intervention Model Description: randomization in two groups: endoscopic ligation or supra-selective embolization and real-life study for a third group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic ligation (Experimental)
  Interventions: Procedure: endoscopic ligation
- Supra-selective embolization (Active Comparator)
  Interventions: Procedure: Supra-selective embolization

INTERVENTIONS:
Procedure: endoscopic ligation — the surgical ligation of one or both sphenopalatine arteries by endoscopic way.
  Arms: endoscopic ligation
Procedure: Supra-selective embolization — occlusion of the terminal branches of the nasal external carotid artery.
  Arms: Supra-selective embolization

SUMMARY:
Current recommendations consider surgical ligation and supra-selective embolization as equivalent in terms of efficacy and there is no clear consensus to choose between one and the other technique. In the absence of medico-economic studies, these recommendations could not be based on any differences in efficiency between the two techniques. The management of patients with severe non-traumatic epistaxis remains controversial and varies according to the hospital and/or university centers. In practice, the use of one or the other technique depends on the habits of each reference center.

DETAILED DESCRIPTION:
The hypothesis is that early ligation of the sphenopalatine arteries would reduce the costs of care for the community while improving the quality of life of patients compared to supra-elective embolization.

This medico-economic superiority could go through:

* reduction in the number of recurrences
* reduction in the length of hospital stays.
* reduction in the cost of postoperative care.
* reduction of iatrogenic complications
* improvement of functional suites upon return home.
* Tertiary prevention of dependency, particularly among the elderly

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe epistaxis who failed treatment with double tamponade for more than 48 hours.
* Patient over 18 years old
* Affiliated patient or beneficiary of a social security scheme.
* Patient accepting the principle of randomization
* Free, informed and written consent, signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patient with epistaxis secondary to facial and/or surgical trauma.
* Patient with epistaxis related to a malignant tumor cause
* Patient with a history of ligation or embolization
* Patient under legal protection and/or curatorship and/or guardianship.
* Impossibility of giving the person informed information and ensuring the subject's compliance due to impaired physical and/or psychological health.
* Patient participating in another research including an exclusion period still in progress
* Pregnant or breastfeeding patient

For non randomized patient

* Patient with a contraindication to general anesthesia: severe and/or decompensated cardiac/hepatic/renal insufficiency, ASA score 4
* Severe hemostasis disorders that cannot benefit from correction.
* History of transient and/or definitive stroke of the ischemic type
* Atheromatous overload

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
incremental cost-utility ratio | Month 18
  the cost-utility ratio integrating direct medical and non-medical costs

SECONDARY OUTCOMES:
number of recurrences | Month 18
time to first recurrence | Month 18
the number of complications | Month 18
nature of complications | Month 18
quality of life with EQ-5D-5L | Month 18
quality of life with SNOT 22 | Month 18
the number of hospitalizations | Month 18
duration of hospitalizations | Month 18
the addiction with KATZ scale | Month 18
incremental cost-effectiveness ratio | Month 18
  the incremental cost-effectiveness ratio (cost/number of recurrences avoided) from the perspective of the community
the description of the costs of care | Month 18
  only for non-randomized patients
financial benefit (1 year) | Month 12
  the annual financial benefit of routine implementation of arterial ligation in the treatment of severe epistaxis, from a community perspective
financial benefit (5 year) | Year 5
  the 5-year financial benefit of routine implementation of arterial ligation in the treatment of severe epistaxis, from a community perspective

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DE BONNECAZE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No